CLINICAL TRIAL: NCT03626337
Title: A Study to Establish a Case Definition of Thiamine Responsive Disorders (TRD) Among Infants in Lao PDR
Brief Title: Thiamine Responsive Disorders (TRD) Among Infants in Lao PDR
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Lao Tropical and Public Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1329444
Record Dates: First submitted 2018-07-17; First posted 2018-08-13 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Thiamine Deficiency
MeSH Terms: conditions — Thiamine Deficiency | interventions — Thiamine; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, plasma and erythrocyte samples will be collected among children. Blood, plasma, erythrocyte and breastmilk samples will be collected among their mothers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital-based cohort: 100 mg thiamine provided via intramuscular and/or intravenous injection (Thiamine 100 MG/ML) daily for 3 days
  Interventions: Drug: Thiamine 100 MG/ML
- Community-based cohort: Sex-, age- and regionally matched comparison group

INTERVENTIONS:
Drug: Thiamine 100 MG/ML — 100 mg thiamine provided as intramuscular injection
  Other Names: Standard of care
  Groups: Hospital-based cohort

SUMMARY:
A hospital- and community-based study in Luang Prabang, Lao PDR, which will include a group of hospitalized children 21 days to <18 months of age who are diagnosed with symptoms compatible with thiamine deficiency disorder (TDD). Based on the infants' response to thiamine administration, children will be defined as either thiamine responsive disorder (TRD) cases or non-responders. A community-based comparison group of infants in the same age range will be included in the study to serve as a control group for identification of potential risk factors.

DETAILED DESCRIPTION:
The study's primary objective is the development of a case definition for TRD among infants and young children with symptoms consistent with TDD, with the case definition being based on those clinical symptoms and other predictors that we find are better able to distinguish those who respond positively to thiamine administration from those who do not respond. As diagnostic tools available to treating physicians may differ by setting, we will repeat analyses after excluding from the set of candidate predictors those that are derived from assessments only available in higher-resource settings, such as laboratory biomarkers and ultrasonography.

A secondary objective is to fill the knowledge gap surrounding biomarkers of thiamine status in at-risk populations. Biomarker cut-offs for TRD will be developed in the hospital cohort and distributions will be characterised in both the hospital and community cohorts. The performance of our proposed cut-off will be compared to the performance of existing literature cut-offs.

Additionally, all identified predictors and biomarker cut-offs will be compared across the community cohort, non-TRD hospital cohort, and TRD hospital cohort to assess the prevalence of risk factors among apparently healthy infants and young children and assess the usefulness of the TRD case definition in various settings.

Infants and children in the target age range, who are seeking care at the collaborating hospital, will be screened by study staff to determine the presence of any of the inclusion criteria. The list of inclusion criteria has been developed based on a broad range of TDD-compatible symptoms to reduce the risk of potentially missing children who would respond clinically to thiamine administration to correct the deficiency. If a child is in the target age range (21 days to <18 months) meets any one of the inclusion criteria, parental consent will be obtained and children will be referred to a study physician for a detailed physical exam. An echocardiogram and cranial ultrasound will be performed to explore the complete range of TDD complications. A venous blood sample will be obtained by venipuncture for assessment of indicators of thiamine status. The data collection will follow a structured timeline after the first thiamine dose has been administered. In particular, the thiamine administration will be defined as hour zero, and the above described physical exam will be repeated 4, 8, 12, 24, 36, 48, and 72 hours after the initial thiamine administration

Blood samples will be analyzed for whole blood thiamine diphosphate (ThDP) and erythrocyte transketolase activity coefficient (ETKac), inflammation and cardiac biomarkers and for a complete blood count (CBC). The purpose of determining these indicators is to better describe the TRD cases and explore differences between TRD cases, non-TRD children and children in the community, with the ultimate goal that these indicators may be useful for screening in the future. Moreover, to determine the association between TRD and maternal thiamine status as a potential risk factor, investigators will collect a blood sample from infants's mothers to assess maternal thiamine status, and among breast feeding mothers a breastmilk sample for assessment of thiamine concentration.

ELIGIBILITY:
Inclusion criteria of hospital-based children:

* 21 days to <18 months and seeking care at the collaborating hospital and meeting at least one of the following inclusion criteria:
* Liver enlargement (>2 cm below right costal margin on calm, supine exam)
* Edema
* Tachypnea (> 60/min for 3-8 wks; >50/min for 2-11 mo; >40/min for 12 - 18 mo)
* Tachycardia (heart rate >160/min for <12 mo; >120/min for 12 mo - 18 mo)
* Oxygen saturation (<92%)
* Difficulty breathing (i.e. chest in-drawing, nasal flaring)
* Refusal to breastfeed or refusal of infant formula or food for greater than 24 hours
* Repetitive or recurring vomiting with no obvious other cause(i.e. vomiting >3 times in past 24 hours)
* Persistent crying not relieved by soothing and feeding with no obvious other cause
* Hoarse voice/cry or loss of voice
* Nystagmus or other unusual eye movement
* Muscle twitching
* Loss of consciousness
* Convulsion
* Opisthotonus / abnormal posturing
* Acute paralysis / flaccid paralysis

Exclusion criteria of hospital-based children:

- None

Inclusion criteria of community-based children, who will be frequency-matched based on sex, age and residence to hospital-based participants :

* Children aged 21 days to <18 months
* Residing in selected communities

Exclusion criteria of community-based children:

- Severe acute illness warranting immediate hospital referral

Inclusion criteria of participants' mothers:

- Mother of hospital-based study participant or community-based study participant

Exclusion criteria of participants' mothers:

* Severe acute illness warranting immediate hospital referral
* Unable to provide informed consent due to reduced decision making ability

Ages: 21 Days to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospitalized children:
  Infants and children in the target age range (21 days to <18 months), who are admitted to the participating hospitals, will be screened by hospital staff to determine the presence of at least one of the inclusion criteria
  Community-based cohort:
  A sex-, age- and regionally-similar comparison group will be enrolled based on the characteristics of the hospitalized group.
  Mothers of all participating infants will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 1394 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Thiamine Responsive Disorder (TRD) | 48-72 hours
  Diagnosis of TRD will be determined based on improvements of initially abnormal physical findings such as hepatomegaly, heart rate, and respiratory rate, and resolution of echocardiographic findings of enlarged and poorly functioning ventricles

SECONDARY OUTCOMES:
Biomarkers of whole blood thiamine diphosphate (ThDP) and erythrocyte transketolase activity coefficient (ETKac) | Baseline
  Associations between ThDP and ETKac with TRD will be determined and appropriate cut-offs of these biomarkers suggesting TRD will be proposed
Hemoglobin and biomarkers of other micronutrients (ferritin, transferrin receptor, retinol binding protein, erythrocyte glutathione reductase activation coefficient (EGRAC)), and inflammation (CRP, AGP) | Baseline
  Nutrition and health status will be assessed to explore potential risk factors for TRD

CONTACTS AND LOCATIONS:
Overall Officials: Sengchanh Kounnavong, MD, PhD, Principal Investigator — Lao Tropical and Public Health Institute
Locations (1):
- Lao Friends Hospital for Children, Luang Prabang, Laos

IPD SHARING:
Plan to Share IPD: Yes
The complete de-identified dataset will be made publically available. Associated data dictionaries will be made available along with the datasets.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 3 years after completion of data collection

REFERENCES:
- [Background] Hess SY, Smith TJ, Fischer PR, Trehan I, Hiffler L, Arnold CD, Sitthideth D, Tancredi DJ, Schick MA, Yeh J, Stein-Wexler R, McBeth CN, Tan X, Nhiacha K, Kounnavong S. Establishing a case definition of thiamine responsive disorders among infants and young children in Lao PDR: protocol for a prospective cohort study. BMJ Open. 2020 Feb 13;10(2):e036539. doi: 10.1136/bmjopen-2019-036539. PMID 32060165
- [Background] Smith TJ, Tan X, Arnold CD, Sitthideth D, Kounnavong S, Hess SY. Traditional prenatal and postpartum food restrictions among women in northern Lao PDR. Matern Child Nutr. 2022 Jan;18(1):e13273. doi: 10.1111/mcn.13273. Epub 2021 Sep 30. PMID 34595830
- [Derived] Hess SY, Arnold CD, Smith TJ, Allen LH, Hampel D, Jones KS, Parkington DA, Meadows SR, Sitthideth D, Kounnavong S. Thiamine Concentration in Human Milk Is Correlated With Maternal and Infant Thiamine Status: A Cross-Sectional Analysis of the Lao Thiamine Study. Matern Child Nutr. 2025 Jul;21(3):e70027. doi: 10.1111/mcn.70027. Epub 2025 Apr 10. PMID 40211576
- [Derived] Hess SY, Smith TJ, Arnold CD, Jones KS, Hampel D, Hiffler L, Trehan I, Fischer PR, Meadows SR, Parkington DA, Brown KH, Sitthideth D, Tan X, Koulman A, Allen LH, Kounnavong S. Assessment of Erythrocyte Transketolase, Whole Blood Thiamine Diphosphate, and Human Milk Thiamine Concentrations to Identify Infants and Young Children Responding Favorably to Therapeutic Thiamine Administration: Findings from the Lao Thiamine Study, a Prospective Cohort Study. Curr Dev Nutr. 2024 May 23;8(6):103786. doi: 10.1016/j.cdnut.2024.103786. eCollection 2024 Jun. PMID 38974350
- [Derived] Smith TJ, Arnold CD, Fischer PR, Trehan I, Hiffler L, Sitthideth D, Stein-Wexler R, Yeh J, Jones KS, Hampel D, Tancredi DJ, Schick MA, McBeth CN, Tan X, Allen LH, Sayasone S, Kounnavong S, Hess SY. A Predictive Model for Thiamine Responsive Disorders Among Infants and Young Children: Results from a Prospective Cohort Study in Lao People's Democratic Republic. J Pediatr. 2024 May;268:113961. doi: 10.1016/j.jpeds.2024.113961. Epub 2024 Feb 17. PMID 38369233
- Available data/document: Statistical Analysis Plan — https://osf.io/jfke3/